CLINICAL TRIAL: NCT05091606
Title: Investigation of Lower and Upper Extremity Perfusion Index (PI) Values in Patients Who Will Have Cesarean Section Under Spinal Anesthesia
Brief Title: Lower and Upper Extremity Perfusion Index (PI) in Pregnant Women Under Spinal Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Collaborators: Mehmet Yilmaz (Unknown)
Responsible Party: Principal Investigator, Ayse KAYHAN, Resident Doctor, Derince Training and Research Hospital
Other Study IDs: DerinceAyşeKayhan1
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Perfusion İndex
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Perfusion İndex in Patients with Spinal Anesthesia — Comparison of lower and upper extremity perfusion index values

SUMMARY:
Spinal anesthesia (SA) is the most preferred method of anesthesia in cesarean deliveries because it eliminates the potential risks associated with airway management in pregnant women. Spinal anesthesia poses a risk of hypotension with an incidence of approximately 70%, resulting from decreased vascular tone due to sympathetic block. Hypotension can cause dizziness in the mother, nausea and vomiting, and acidosis in the fetus. Therefore, the prevention and treatment of postspinal hypotension has been an important area of research in obstetric anesthesia.

The Perfusion Index (PI) is the ratio of pulsatile blood flow (arterial chamber) to non-pulsatile static blood flow (venous and capillaries) in a patient's peripheral tissue, such as the fingertip, toe, or earlobe. This can be obtained from a pulse oximeter. This is non-invasive and continuous monitoring.

The pulse variability index (PVI) represents changes in PI that occur during one or more complete respiratory cycles. PVI is found by calculating over PI changes. Allows evaluation of intravascular volume; and a higher PVI is associated with greater responsiveness to fluid volumes.

In our work; We will simultaneously observe PI and PVI changes in the lower and upper extremities in the study group patients. When we look at the previous studies; we see that the parameters (PI and PVI) that we will look at are evaluated with different combinations in our study group patients. When we look at these studies again; We saw that contradictory results were obtained for the same parameters.

In our study, patients will be verbally informed in detail about the study in the preoperative period and their consent will be obtained. While the patients are taken to the operating room and monitored, the saturation probe will be connected to the 2nd finger of the upper and lower extremities of the patients, and the PI and PVI values in both extremities will be measured simultaneously. PI and PVI values and vital values (SAB, MAP, HR, SPO2) in both extremities before spinal anesthesia; intraoperative SAP, MAP, HR, SPO2, ephedrine requirement, atropine requirement and PI and PVI values in both extremities will be recorded.

As a result; In our study, we aimed to observe simultaneous changes in PI and PVI in the lower and upper extremities in pregnant patients who will undergo cesarean section under spinal anesthesia, which is our study group.

ELIGIBILITY:
Inclusion Criteria:

* ASA1 and ASA2 patients
* Patients over the age of 18
* Patients suitable for spinal anesthesia
* Patients who agreed to participate in the study with informed consent
* Patients who will have an elective cesarean section

Exclusion Criteria:

* ASA3 and ASA4 patients
* Patients younger than 18 years old
* Patients for whom spinal anesthesia is contraindicated
* Patients who are hemodynamically unstable
* Patients to be taken to emergency cesarean section
* Patients with drug allergies
* Patients with finger deformities that prevent the insertion of the saturation probe
* Patients who did not agree to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA 1-2 patients over the age of 18 who have undergone elective cesarean section and accept spinal anesthesia will be included.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Is there any difference between upper and lower extremitiy perfusion index values? | 4 months
  Observation of PI values in cesarean sections under spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)